CLINICAL TRIAL: NCT03906006
Title: A Single-Center, Randomized, Double-Blind, Placebo-Controlled Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Ascending Oral Doses of ABP-671 in Healthy Volunteers in the United States
Brief Title: A Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ABP-671 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atom Therapeutics Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABP-671-101
Record Dates: First submitted 2019-04-04; First posted 2019-04-08 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Gout; Hyperuricemia
Keywords: gout; hyperuricemia
MeSH Terms: conditions — Gout; Hyperuricemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- ABP-671, Cohort 1- (Experimental): ABP-671, Cohort 1 participants received 50 mg ABP-671 single agent or placebo during dose escalation (6 active: 2 placebo).
  Interventions: Drug: ABP-671; Other: Placebo
- ABP-671, Cohort 2- (Experimental): ABP-671, Cohort 2 participants will receive 0.1 mg ABP-671 single agent or placebo during dose escalation (6 active: 2 placebo).
  Interventions: Drug: ABP-671; Other: Placebo
- ABP-671, Cohort 3- (Experimental): ABP-671, Cohort 3 participants will receive 0.5 mg ABP-671 single agent or placebo during dose escalation (6 active: 2 placebo).
  Interventions: Drug: ABP-671; Other: Placebo
- ABP-671, Cohort 4- (Experimental): ABP-671, Cohort 4 participants will receive 1.0 mg ABP-671 single agent or placebo during dose escalation (6 active: 2 placebo).
  Interventions: Drug: ABP-671; Other: Placebo

INTERVENTIONS:
Drug: ABP-671 — Drug: ABP-671, single oral dose
Other: Placebo — Other: Placebo, single oral dose

SUMMARY:
The purpose of this study is to assess the safety, tolerability, pharmacokinetics and pharmacodynamics of single ascending doses of ABP-671 administered orally in healthy volunteers.

DETAILED DESCRIPTION:
Primary Objectives:

• To assess the safety and tolerability of single ascending oral doses of ABP-671 in Healthy Volunteers (HVs).

Secondary Objectives:

• To characterize the pharmacokinetics (PK) and pharmacodynamics (PD) profiles of single ascending oral doses of ABP-671 in HVs.

ELIGIBILITY:
Inclusion Criteria

1. Healthy (no clinically significant health concerns), as determined by medical history, physical examination, 12-lead ECG, and vital signs.
2. Participants serum uric acid level at screening ≥ 4.0 mg/dL to ≤ 5.5 mg/dL for males, and ≥ 4.0 mg/dL to ≤ 5.0 mg/dL for females.
3. Participants must have a body mass index (BMI) between 18 and 32 kg/m2 and a body weight of 50 kg or higher.
4. Participants must have normal blood chemistry or results considered not clinically significant by the investigator including electrolytes, alkaline phosphatase, total protein, albumin, aspartate aminotransferase (AST), alanine aminotransferase (ALT), total bilirubin, uric acid, creatinine, blood urea nitrogen (BUN), and glucose at Screening Visit and at Pre-dose Visit.
5. Participants are able to understand the study procedures and risks involved and must provide signed informed consent to participate in the study.

Exclusion Criteria

1. Participants with any history or clinical manifestations of significant metabolic, hematological, pulmonary, including latent tuberculosis, cardiovascular, gastrointestinal including cholecystectomy, neurologic, hepatic, renal, urological, or psychiatric disorders.
2. Participants who have any history or suspicion of kidney stones.
3. Participants who have used prescription drugs, over-the-counter drugs, or herbal remedies within 14 days before Day 1 of study medication dosing. Females who have received hormone replacement therapy (HRT) within 28 days prior to dosing.
4. Women who are pregnant or breastfeeding.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2018-10-17 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-06-20 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | baseline to 7 days
  Incidence of adverse events
Maximum tolerable dose | baseline to 7 days
  Maximum tolerable dose

SECONDARY OUTCOMES:
Peak plasma concentration | baseline to 72 hours
  Peak plasma concentration
half-life | baseline to 72 hours
  half-life
area under the curve | baseline to 72 hours
  area under the curve
volume of distribution | baseline to 72 hours
  volume of distribution
level of serum and urine uric acid | baseline to 72 hours
  level of serum and urine uric acid
level of serum and urine creatinine | baseline to 72 hours
  level of serum and urine creatinine

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Armas, M.D., Principal Investigator — Celerion
Locations (1):
- Celerion, Tempe, Arizona, United States